CLINICAL TRIAL: NCT04240470
Title: Endovascular Stroke Treatment Only (ESTO) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Eskisehir Osmangazi University Training and Research Hospital (Unknown); Kartal Dr. Lütfi Kirdar City Hospital (Unknown); Sakarya University Training and Research Hospital (Unknown); Ondokuz Mayis University Training and Research Hospital (Unknown)
Responsible Party: Principal Investigator, Adnan Qureshi, Professor of Neurology, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019141
Record Dates: First submitted 2020-01-13; First posted 2020-01-27 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; endovascular treatment; recombinant tissue plasminogen activator; mechanical thrombectomy
MeSH Terms: conditions — Ischemic Stroke | interventions — Thrombectomy

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to receive endovascular treatment for acute ischemic stroke (mechanical thrombectomy) alone without using IV rt-PA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thrombectomy (Experimental): Participants will receive endovascular treatment (mechanical thrombectomy) alone without using IV rt-PA.
  Interventions: Procedure: Thrombectomy

INTERVENTIONS:
Procedure: Thrombectomy — Participants will receive endovascular treatment (mechanical thrombectomy) alone without using IV rt-PA.

SUMMARY:
The specific aims of this study are to:

1. Determine whether the endovascular treatment (mechanical thrombectomy) alone without using intravenous (IV) recombinant tissue plasminogen activator (rt-PA) in acute ischemic stroke patients demonstrates "promise" or a lack thereof ("futility") in deciding what would be the next phase III trial.
2. Determine the proportion of subjects with slight or no disability (a modified Rankin score (mRS) of 0-2) at 3 months after receiving endovascular treatment (mechanical thrombectomy) alone without using IV rt-PA and compare with historical controls who were treated with IV rt-PA to identify (or lack of) futility.
3. Determine the proportion of subjects with improvement in the National Institutes of Health Stroke Scale (NIHSS) score of ≥8 points or achieving a score of 0-1 at 24 hours after the onset of stroke among subjects with acute ischemic stroke after receiving endovascular treatment (mechanical thrombectomy) alone without using IV rt-PA.
4. Determine the proportion of subjects with angiographic recanalization on post procedure angiogram according to modified Thrombolysis in Cerebral Infarction (TICI) perfusion flow categories among subjects with acute ischemic stroke after receiving endovascular treatment (mechanical thrombectomy) alone without using IV rt-PA.
5. Determine the proportion of subjects with treatment-related serious adverse events (SAEs) within 72 hours and development of symptomatic intracranial hemorrhage at 27 ±3hrs post treatment among subjects with acute ischemic stroke after receiving endovascular treatment (mechanical thrombectomy) alone without using IV rt-PA.

DETAILED DESCRIPTION:
A phase II trial is proposed to address the question whether administration of intravenous (IV) recombinant tissue plasminogen activator (rt-PA) in acute ischemic stroke patients who are candidates for endovascular treatment provides any additional value. The phase II trial will treat consecutive patients who are candidates for IV rt-PA and mechanical thrombectomy with just mechanical thrombectomy alone. Such trial will generate the necessary data for a definitive phase III trial. The trial is designed based on low rate of recanalization in patients with major arterial occlusion with IV rt-PA alone and no difference in rate of recanalization or distal embolization in patients who receive IV rt-PA and those who do not prior to mechanical thrombectomy. The rates of intracranial hemorrhage (ICH) and cost of hospitalization are higher when IV rt-PA is administered prior to mechanical thrombectomy. The trial will determine the proportion of patients with slight or no disability (a modified Rankin score (mRS) of 0-2) at 3 months after receiving endovascular treatment (mechanical thrombectomy) alone without using IV rt-PA and compare with historical controls who were treated with IV rt-PA to determine futility.

ELIGIBILITY:
Inclusion Criteria:

* • Age: 18 through 90 years (i.e., candidates must have had their 18th birthday, but not had their 91st birthday).

  * Symptom onset within 4.5 hours of onset of stroke symptoms. Time of onset is defined as the last time when the patient was witnessed to be at baseline (i.e., subjects who have stroke symptoms upon awakening will be considered to have their onset at beginning of sleep).
  * An NIHSS ≥ 6 at the time of evaluation. Thrombolysis in Cerebral Infarction (TICI) 0-1 flow in the intracranial internal carotid artery, M1 or M2 segment of the middle cerebral artery (MCA), or carotid terminus confirmed by Computed Tomography (CT) or magnetic resonance (MR) angiography that is accessible to the stent retriever or suction thrombectomy catheter.
  * The procedure can be initiated according to guidelines of AHA/ASA which state that the treatment should be initiated (groin puncture) within 6 hours of symptom onset.

Exclusion Criteria:

* Clinical Exclusion Criteria

  * History of stroke in the past 3 months.
  * Previous intracranial hemorrhage, intracranial neoplasm, subarachnoid hemorrhage, or ruptured brain arteriovenous malformation.
  * Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT scan is normal.
  * Severe hypertension at time of treatment; systolic blood pressure > 185 or diastolic > 110 mm Hg that cannot be corrected prior to treatment.
  * Presumed septic embolus.
  * Major surgery within the previous 14 days.
  * Recent (within 90 days) severe head trauma or head trauma with loss of consciousness.
  * Gastrointestinal malignancy or gastrointestinal hemorrhage within 21 days.
  * Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; or oral anticoagulant therapy with International Normalized Ratio (INR) > 1.7 or institutionally equivalent prothrombin time or platelets count <100,000 per microliter.
  * Women of childbearing potential who are known to be pregnant and/or lactating or who have positive pregnancy tests on admission.
  * Patients with renal failure that require hemodialysis or peritoneal dialysis.
  * Low molecular weight heparins (such as Dalteparin, Enoxaparin, Tinzaparin, Fondaparinux) as deep vein thrombosis (DVT) prophylaxis or in full dose within the last 24 hours from screening unless anti-activated factor X (anti-factor Xa) assay less than 200% of control value.
  * Patients who have received heparin within 48 hours must have a normal partial thromboplastin time (PTT) to be eligible.
  * Patients who have received heparin or a direct thrombin inhibitor (Angiomax, Argatroban, Refludan) must have a normal PTT to be eligible.
  * Patients on dabigatran etexilate mesylate (Pradaxa), rivaroxaban (Xarelto), apixaban (Eliquis), and edoxaban (Savaysa) may be considered after 48 hours after last intake of medication in patients with normal renal function (CrCl > 60 mL/minute). If moderate renal impairment, CrCl of 30-59 mL/minute, last dose should be 72 hours before procedure and 96 hours in severe renal impaired patients (CrCl of 15-29 mL/minute). The time interval between the last dose administration and the neurointerventional procedure appears to be the most reliable criterion for assessing the risk of bleeding events. Patients in whom time of last dose ingestion is unknown or within last 48 hours, can be included under following circumstances: normal PTT for dabigatran, normal prothrombin time for rivaroxaban, or anti-activated factor X (anti-factor Xa) assay rivaroxaban (Xarelto), apixaban (Eliquis), or edoxaban (Savaysa) less than 200% of control value.
  * Subjects with an arterial puncture at a non-compressible site or a lumbar puncture in the previous 7 days.
  * Patients with a seizure at onset of stroke.
  * Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations.
  * Other serious, advanced, or terminal illness.
  * Current participation in another research drug treatment protocol (patient cannot start another experimental agent until after 90 days).

Informed consent is not or cannot be obtained. For example, obtunded patients are not automatically excluded from the study. However, if the next of kin or legal guardian (i.e., the individual legally empowered in the state where the consent is obtained) cannot provide consent, randomization and entry into the study could not proceed.

CT Scan Exclusion Criteria

* High density lesion consistent with hemorrhage of any degree.
* Significant mass effect with midline shift.
* Large (more than 1/3 of the middle cerebral artery) regions of clear hypodensity on the baseline CT scan or ASPECTS of < 4.
* Sulcal effacement and / or loss of grey-white differentiation alone are not contraindications for treatment.

CT Angiographic Exclusion Criteria

* Angiographic evidence of carotid dissection or complete cervical carotid occlusion.
* Arterial tortuosity, calcification, pre-existing stent, and/or stenosis, which would prevent the thrombectomy device from reaching the target vessel and/or preclude safe recovery of the endovascular devices.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-23 (Actual); Study Completion 2021-10-23 (Actual)

PRIMARY OUTCOMES:
Favorable Outcome | 90 days
  Modified Rankin Scale (mRS) score of 0-2: 0, No symptoms at all; 1, No significant disability despite symptoms; able to carry out all usual duties and activities; 2, Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance. The modified Rankin Scale score ranges from 0, indicating no symptoms, to 6, indicating death.

SECONDARY OUTCOMES:
Angiographic Recanalization | Within 6 hours of interventional treatment
  Post procedure angiogram according to modified Thrombolysis in Cerebral Infarction perfusion flow categories:
  0 = No perfusion. No antegrade flow beyond the point of occlusion.
  1. = Perfusion past the initial obstruction but limited distal branch filling with little or slow distal perfusion
  2. A = Perfusion of less than half of the vascular distribution of the occluded artery (eg, filling and perfusion through 1 M2 division)
  2B = Perfusion of half or greater of the vascular distribution of the occluded artery (eg, filling and perfusion through 2 or more M2 divisions) 3 = Full perfusion with filling of all distal branches perfusion flow categories
Early Neurological Improvement | 24 hours post enrollment
  National Institutes of Health Stroke Scale (NIHSS) score of ≥8 points or achieving a score of 0-1 at 24 hours after the onset of stroke. NIHSS quantifies neurologic deficits in 11 categories. Level of consciousness, horizontal eye movement, visual fields, facial palsy, movement in each limb, sensation, language & speech, and extinction or inattention on one side of the body are tested. Scores range from 0 to 42, with 0 indicating normal function and higher scores indicating greater deficit severity.
Quality of Life Status Using Standardized EQ-5D-3L (EuroQol Five Dimension, Three-Level) Questionnaire. | 90 days
  The EQ-5D-3L questionnaire consists of 5 questions in 5 different domains and allows for responses from 1 (the best outcome) to 3 (the worst outcome) in each of five categories (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Total scores range from 5 to 15, with lower scores indicating better quality of life and a higher score indicating a worse quality of life.
Quality of Life Status Using EQ VAS (EuroQol Visual Analog Scale) Scores. | 90 days
  EuroQol outcome measurements is a printed 20 cm visual analogue scale (EQ VAS) that appears somewhat like a thermometer, on which a score from 0 (worst imaginable health state or death) to 100 (best imaginable health state) is marked by the patient (or, when necessary, their proxy) with the scale in view.

OTHER OUTCOMES:
Treatment-Related Serious Adverse Events | Within 72 hours of interventional treatment
  Assessement by the investigators for all patients
Symptomatic intracranial hemorrhage | 24 ± 3hrs post enrollment
  Any hematoma within ischemic field with some mild space occupying effect but involving ≤ 30% of the infarcted area, hematoma within ischemic field with space-occupying effect involving >30% of the infarcted area, any intraparenchymal hemorrhage remote from the ischemic field, subarachnoid hemorrhage, or intraventricular hemorrhage associated with a 4 points or more worsening on the NIHSS within 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Qureshi, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No